CLINICAL TRIAL: NCT05520320
Title: Assessment of Long-term Outcomes After Transplantation of Donor Livers Preserved by Hypothermic Oxygenated Machine Perfusion (HOPE): a Retrospective Cohort Analysis of Real-world Data (IDEAL-D Stage 4)
Brief Title: Long-term Outcomes After Hypothermic Oxygenated Machine Perfusion of Donor Livers Using Real-world Data
Acronym: HOPE-REAL
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: HOPE-REAL study
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Organ Preservation; Liver Transplantation; Hypothermic Machine Perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hypothermic oxygenated machine perfusion (any device) — After static cold storage, all grafts included in this study are subjected to >1 hour of hypothermic oxygenated machine perfusion at 4-12°C with an acellular perfusion solution.

SUMMARY:
End-ischemic hypothermic oxygenated machine perfusion (HOPE) of human donor livers mitigates ischemia-reperfusion injury, resulting in a reduction of post-reperfusion syndrome, early allograft dysfunction and biliary complications, when compared with static cold storage. According to IDEAL-D (Idea, Development, Exploration, Assessment, Long term study-Framework for Devices), with several published randomized controlled trials on short-to-medium term outcomes, scientific evidence for HOPE has currently reached stage 3. Assessment of long-term outcomes after HOPE preservation based on real-world data (i.e., IDEAL-D stage 4) is currently still lacking. Therefore, we aim to conduct an international, multi-center, retrospective, observational cohort study to assess long-term outcomes after transplantation of donor livers preserved by hypothermic oxygenated machine perfusion (HOPE).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) who underwent liver transplantation of donor livers preserved with end-ischemic HOPE (including donation after normothermic regional perfusion) between 01.01.2012 and 31.12.2021.

Exclusion Criteria:

* Simultaneous multiorgan transplantations, sequential normothermic machine perfusion (e.g., DHOPE-COR-NMP, but not NRP), living partial liver donation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) undergoing liver transplantation of donor livers preserved with end-ischemic HOPE.
Sampling Method: Non-Probability Sample
Enrollment: 1202 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Death-censored graft survival, assessed by survival analysis methods | Up to 5-years
  Defined as time from liver transplantation until re-transplantation or death due to graft dysfunction

SECONDARY OUTCOMES:
Overall graft survival | Up to 5-years
  Defined as time from liver transplantation until re-transplantation or all-cause death
Overall patient survival | Up to 5-years
  Defined as time from liver transplantation until all-cause death
Arterial and biliary complication-free survival (ABCFS) | Up to 5-years
  Defined as time from liver transplantation until occurrence of an arterial or biliary complication of Dindo-Clavien grade ≥3, dated at the time of interventional, endoscopic, or surgical treatment required to correct it (Savier E, De Rycke Y, Lim C, et al. Novel Composite Endpoint for Assessing Outcomes in Liver Transplantation: Arterial and Biliary Complication-Free Survival. Liver Transpl. 2022;28(1):75-87. doi:10.1002/lt.26269)
Incidence of biliary complications | Up to 5-years
  Defined as a composite of:
  * Non-anastomotic biliary strictures: any irregularity or narrowing of the lumen of the intrahepatic or extrahepatic donor bile ducts, excluding the biliary anastomosis, diagnosed with the use of cholangiography in combination with clinical symptoms (e.g., jaundice or cholangitis) or an elevation of cholestatic laboratory variables, in the presence of a patent hepatic artery
  * Anastomotic biliary strictures: strictures occurring at the anastomosis of donor choledochal duct and recipient choledochal duct or jejunal Roux-limb
  * Biliary leakage: fluid with an elevated (>3x serum) bilirubin level in the abdominal drain or intra-abdominal fluid on or after post-operative day 3 or the need for radiological intervention (i.e. interventional drainage) owing to biliary collections or re-laparotomy due to biliary peritonitis
Incidence of vascular complications | Up to 5-years
  Defined as a composite of:
  * Hepatic arterial thrombosis: radiologically or surgically proven thrombosis of the hepatic artery
  * Portal vein thrombosis: radiologically or surgically proven thrombosis of the portal vein
  * Venous outflow tract obstruction: radiologically or surgically proven thrombosis of the main hepatic veins or the inferior vena cava
Incidence of acute cellular rejection | Up to 5-years
  Defined as biopsy proven Banff grade 2 or 3 rejection (Demetris AJ, Bellamy C, Hübscher SG, et al. 2016 Comprehensive Update of the Banff Working Group on Liver Allograft Pathology: Introduction of Antibody-Mediated Rejection. Am J Transplant. 2016;16(10):2816-2835. doi:10.1111/ajt.13909)
Incidence of chronic rejection | Up to 5-years
  Defined as histopathological evidence of immunologic injury with irreversible damage to the bile ducts, arteries, and veins (Demetris A, Adams D, Bellamy C, et al. Update of the International Banff Schema for Liver Allograft Rejection: working recommendations for the histopathologic staging and reporting of chronic rejection. An International Panel. Hepatology. 2000;31(3):792-799. doi:10.1002/hep.510310337)
Incidence of re-transplantation | Up to 5-years
  Defined as proportion of patients who underwent liver re-transplantation for any cause
Incidence of recurrence of primary disease (including recurrence of malignancies) | Up to 5-years
  Defined as histological or radiologically confirmed recurrence
Incidence of new-onset chronic kidney disease | Up to 5-years
  Defined as renal impairment (kidney morphology, pathology, imaging, blood or urine composition abnormalities) persisting for >3 months with or without eGFR decrease, and/or eGFR <60 for >3 months with or without renal impairment (Levey AS, Eckardt K-U, Tsukamoto Y, et al. Definition and Classification of Chronic Kidney Disease: A Position Statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x)
Incidence of new-onset diabetes after transplantation | Up to 5-years
  Defined as symptoms of diabetes plus casual plasma glucose levels ≥200 mg/dL (11.1 mmol/L) or fasting plasma glucose ≥126 mg/dL (7.0 mmol/L) or 2 hours plasma glucose ≥200 mg/dL (11.1 mmol/L during an oral glucose tolerance testing (Davidson J, Wilkinson A, Dantal J, et al. New-onset diabetes after transplantation: 2003 International consensus guidelines. Proceedings of an international expert panel meeting. Barcelona, Spain, 19 February 2003. Transplantation. 2003;75(10 Suppl):SS3-24. doi:10.1097/01.TP.0000069952.49242.3E)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent E de Meijer, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- University Medical Center Groningen, Groningen, Netherlands
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eden J, Bruggenwirth IMA, Berlakovich G, Buchholz BM, Botea F, Camagni S, Cescon M, Cillo U, Colli F, Compagnon P, De Carlis LG, De Carlis R, Di Benedetto F, Dingfelder J, Diogo D, Dondossola D, Drefs M, Fronek J, Germinario G, Gringeri E, Gyori G, Kocik M, Kucukerbil EH, Koliogiannis D, Lam HD, Lurje G, Magistri P, Monbaliu D, Moumni ME, Patrono D, Polak WG, Ravaioli M, Rayar M, Romagnoli R, Sorensen G, Uluk D, Schlegel A, Porte RJ, Dutkowski P, de Meijer VE. Long-term outcomes after hypothermic oxygenated machine perfusion and transplantation of 1,202 donor livers in a real-world setting (HOPE-REAL study). J Hepatol. 2025 Jan;82(1):97-106. doi: 10.1016/j.jhep.2024.06.035. Epub 2024 Jul 3. PMID 38969242